CLINICAL TRIAL: NCT04912063
Title: A Phase 1b Dose Escalation Study of Lemzoparlimab in Combination With Venetoclax and/or Azacitidine in Subjects With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Study to Evaluate Adverse Events and Movement of Lemzoparlimab in Body When Used Intravenously (IV) With Azacitidine Subcutaneously or IV and Venetoclax Orally in Participants With Acute Myeloid Leukemia and With Azacitidine With or Without Venetoclax in Participants With Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-866; 2021-000514-41 (EudraCT Number)
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Lemzoparlimab; TJ011133; ABBV-IMAB-TJC4; Venetoclax; ABT-199; GDC-0199; VENCLEXTA; VENCLYXTO; Azacitidine; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasms | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Lemzoparlimab + Azacitidine + Venetoclax in AML (Escalation) (Experimental): Lemzoparlimab (TJ011133) co-administered with azacitidine and venetoclax in escalated doses in participants with treatment-naïve acute myeloid leukemia (AML) who are ineligible for standard induction therapy.
  Interventions: Drug: Lemzoparlimab; Drug: Azacitidine; Drug: Venetoclax
- Lemzoparlimab + Azacitidine + Venetoclax in MDS (Escalation) (Experimental): Lemzoparlimab (TJ011133) co-administered with azacitidine and venetoclax in escalated doses in participants with treatment-naïve higher-risk myelodysplastic syndrome (MDS).
  Interventions: Drug: Lemzoparlimab; Drug: Azacitidine; Drug: Venetoclax
- Lemzoparlimab + Azacitidine in MDS (Escalation) (Experimental): Lemzoparlimab (TJ011133) co-administered with azacitidine in escalated doses in participants with treatment-naïve higher-risk myelodysplastic syndrome (MDS).
  Interventions: Drug: Lemzoparlimab; Drug: Azacitidine
- Lemzoparlimab + Azacitidine + Venetoclax in AML (Expansion) (Experimental): Lemzoparlimab (TJ011133) co-administered with azacitidine and venetoclax in expansion cohort in participants with treatment-naïve acute myeloid leukemia (AML) who are ineligible for standard induction therapy.
  Interventions: Drug: Lemzoparlimab; Drug: Azacitidine; Drug: Venetoclax
- Lemzoparlimab + Azacitidine + Venetoclax in MDS (Expansion) (Experimental): Lemzoparlimab (TJ011133) co-administered with azacitidine and venetoclax in expansion cohort in participants with treatment-naïve higher-risk myelodysplastic syndrome (MDS).
  Interventions: Drug: Lemzoparlimab; Drug: Azacitidine; Drug: Venetoclax
- Lemzoparlimab Monotherapy in AML (Japan Only Escalation) (Experimental): Lemzoparlimab (TJ011133) administered in escalated doses in participants with treatment-naïve acute myeloid leukemia (AML) who are ineligible for standard induction therapy.
  Interventions: Drug: Lemzoparlimab
- Lemzoparlimab Monotherapy in MDS (Japan Only Escalation) (Experimental): Lemzoparlimab (TJ011133) administered in escalated doses in participants with treatment-naïve higher-risk myelodysplastic syndrome (MDS).
  Interventions: Drug: Lemzoparlimab

INTERVENTIONS:
Drug: Lemzoparlimab — Intravenous (IV) Infusion
  Other Names: TJ011133; ABBV-IMAB-TJC4
Drug: Azacitidine — Subcutaneous Injection or Intravenous (IV) Injection/Infusion
  Arms: Lemzoparlimab + Azacitidine + Venetoclax in AML (Escalation); Lemzoparlimab + Azacitidine + Venetoclax in AML (Expansion); Lemzoparlimab + Azacitidine + Venetoclax in MDS (Escalation); Lemzoparlimab + Azacitidine + Venetoclax in MDS (Expansion); Lemzoparlimab + Azacitidine in MDS (Escalation)
Drug: Venetoclax — Oral Tablet
  Other Names: Venclexta; Venclyxto; ABT-199; GDC-0199
  Arms: Lemzoparlimab + Azacitidine + Venetoclax in AML (Escalation); Lemzoparlimab + Azacitidine + Venetoclax in AML (Expansion); Lemzoparlimab + Azacitidine + Venetoclax in MDS (Escalation); Lemzoparlimab + Azacitidine + Venetoclax in MDS (Expansion)

SUMMARY:
Acute myeloid leukemia (AML) is one of the most aggressive blood cancers, with a very low survival rate and few options for participants who are unable to undergo intensive chemotherapy, the current standard of care. This study is to evaluate how safe lemzoparlimab is and how it moves within the body when used along with azacitidine and/or venetoclax in adult participants with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS). Adverse events and maximum tolerated dose (MTD) of lemzoparlimab will be assessed.

Lemzoparlimab (TJ011133) is being evaluated in combination with azacitidine and venetoclax for the treatment of acute myeloid leukemia (AML) and with azacitidine with/without venetoclax for myelodysplastic syndrome (MDS). Study doctors place the participants in 1 of 5 groups, called treatment arms. Each group receives a different treatment. Adult participants with a diagnosis of AML or MDS will be enrolled. Around 80 participants will be enrolled in the study in approximately 50 sites worldwide.

Participants will receive lemzoparlimab (IV) once weekly (Q1W), venetoclax oral tablets once daily (QD) for 28 days (AML participants) or 14 days (MDS participants) and Azacitidine by SC or IV route QD for 7 days of each 28-day cycle.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented confirmation of acute myeloid leukemia (AML) according to the World Health Organization (WHO) criteria, previously untreated [OR]
* Documented diagnosis of previously untreated de novo myelodysplastic syndrome (MDS) according to the 2017 WHO classification with presence of < 20% bone marrow blasts per marrow biopsy/aspirate.
* Participants with documented MDS must meet the following disease activity criteria:

  * Overall revised international prognostic scoring system (IPSS-R) score > 3 (intermediate, high, or very high);
  * Eastern cooperative oncology group (ECOG) performance status of 0 to 2;
  * Hematopoietic stem cell transplant (HSCT) ineligible, or participant who chooses not to undergo HSCT.
* Participants with documented AML with adverse cytogenetic and/or molecular risk, and must be considered ineligible for induction therapy defined by the following:

  * >= 75 years of age; [OR]
  * >= 18 to 74 years of age with at least one of the following comorbidities: --- Eastern cooperative oncology group (ECOG) performance status of 2 to 3; --- Cardiac history of congestive heart failure requiring treatment or ejection fraction <= 50% or chronic stable angina;

    * Diffusion capacity of lung (DLCO) <= 65% or forced expiratory volume during the first second (FEV1) <= 65%;
    * Creatinine clearance >= 30 mL/min to < 45 mL/min;
    * Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × upper limit of normal (ULN);
    * Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy or the participant declines to receive intensive chemotherapy.

Japan Safety Lead-In Phase:

* Documented confirmation of AML according to WHO criteria, relapsed or refractory (R/R) disease without other standard of care treatments.
* Documented diagnosis of MDS according to the 2017 WHO classification with presence of < 20% bone marrow blasts per marrow biopsy/aspirate, with intermediate- and high-risk relapsed/refractory MDS.
* Documented MDS must meet the following disease activity criteria:

  * ECOG performance status of 0 to 2.

Exclusion Criteria:

* Participants with documented AML with acute promyelocytic leukemia and considered eligible for induction therapy.
* Participant with documented AML having prior diagnosis of:

  -- known active central nervous system involvement with AML.
* Participants with documented MDS having prior diagnosis of:

  * MDS evolving from a pre-existing myeloproliferative neoplasm (MPN);
  * MDS/MPN including chronic myelomonocytic leukemia, atypical chronic myeloid leukemia, juvenile myelomonocytic leukemia and unclassifiable MDS/MPN.
* History of allogeneic HSCT or solid organ transplantation.
* Previous exposure to anti-CD47 therapies.
* History of an active malignancy within the past 2 years prior to Screening, with the exception of:

  -- Adequately treated carcinoma in situ of the cervix uteri or carcinoma in situ of the breast;
  * Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin;
  * Asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Conditions that could interfere with drug absorption including but not limited to short bowel syndrome.

Japan Safety Lead-In Phase:

* Documented AML have Acute Promyelocytic Leukemia.
* Participant with documented AML having prior diagnosis of:

  -- Chronic myeloid leukemia with or without BCR-ABL1 translocation and AML with BCR-ABL1 translocation.
* Participants with documented MDS having prior diagnosis of:

  * Therapy-related MDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) of Lemzoparlimab (TJ011133) When Co-administered With Venetoclax and Azacitidine in Participants With Treatment-Naïve Acute Myeloid Leukemia (AML) Ineligible for Standard Induction Therapy | Up to 30 days after first dose of study drug
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications and occurring during the first 4 weeks after administration of the first dose and that meets additional criteria as described in the protocol.
DLTs of Lemzoparlimab (TJ011133) When Co-administered With Azacitidine With or Without Venetoclax in Participants With Treatment-Naïve Higher-Risk Myelodysplastic Syndrome (MDS) | Up to 30 days after first dose of study drug
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications and occurring during the first 4 weeks after administration of the first dose and that meets additional criteria as described in the protocol.
Dose Limiting Toxicities (DLTs) of Lemzoparlimab (TJ011133) as a Monotherapy in Japanese Participants with Relapsed/Refractory (R/R) AML | Up to 30 days after first dose of study drug
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications and occurring during the first 4 weeks after administration of the first dose and that meets additional criteria as described in the protocol.
DLTs of Lemzoparlimab (TJ011133) as a Monotherapy in Japanese Participants with R/R MDS | Up to 30 days after first dose of study drug
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications and occurring during the first 4 weeks after administration of the first dose and that meets additional criteria as described in the protocol.

SECONDARY OUTCOMES:
Best Overall Response of Complete Remission (CR) for AML | Up to approximately 3 years
  Best overall response of complete remission (CR), defined as achieving CR according to modified international working group (IWG) 2003 criteria for AML.
Best Overall Response of Composite CR (CRc) for AML | Up to approximately 3 years
  Best overall response of composite CR (CRc), [CR or CR with incomplete blood count recovery (CRi)] according to modified IWG 2003 criteria for AML.
Best Overall Response of CR or Complete Remission With Partial Hematologic Recovery (CRh) for AML | Up to approximately 3 years
  Best overall response of CR or CRh, defined according to modified IWG 2003 criteria for AML.
Duration of Response (DOR) for AML | Up to approximately 3 years
  Duration of response (DOR), defined for participants who achieve a best overall response, as the time from the first occurrence of response to disease progression/relapse from CR, CRi or CRh or death from disease progression, whichever occurs first.
Event-Free Survival (EFS) for AML | Up to approximately 3 years
  Event-free survival (EFS), defined as time from first dose of any study drug (lemzoparlimab or venetoclax or azacitidine) to the date of progressive disease (PD), relapse from CR or CRi, treatment failure defined as failure to achieve CR, CRi or MLFS after at least 6 cycles of study treatment, or death from any cause, whichever occurs first.
Overall Survival (OS ) for AML | Up to approximately 3 years
  Overall survival (OS), defined as the time from the date of the first dose of any study drug (lemzoparlimab or venetoclax or azacitidine) to death from any cause.
Best Overall Response of CR, for MDS | Up to approximately 3 years
  Best overall response of CR per the modified IWG 2006 criteria for MDS.
Best Overall Response of Marrow-Complete Remission (mCR), for MDS | Up to approximately 3 years
  Best overall response of marrow-complete remission (mCR), per the modified IWG 2006 criteria for MDS.
Best Overall Response of CR or PR for MDS | Up to approximately 3 years
  Best overall response of CR or PR, per the modified IWG 2006 criteria for MDS.
Best Overall Response of CR or PR or mCR, for MDS | Up to approximately 3 years
  Best overall response of CR or PR or mCR, per the modified IWG 2006 criteria for MDS.
Hematologic Improvement (HI), for MDS | Up to approximately 3 years
  Hematologic improvement (HI), defined as a participant achieving erythroid/platelet/neutrophil responses.
Red Blood Cell Transfusion Independence (TI), for MDS | Up to approximately 3 years
  Red blood cell transfusion independence (TI), defined as a participant who is transfusion dependent at baseline achieved TI post-baseline.
Platelet TI, for MDS | Up to approximately 3 years
  Platelet TI, defined as a participant who is transfusion dependent at baseline achieved TI post-baseline.
DOR, for MDS | Up to approximately 3 years
  DOR, defined for participants who achieve a best overall response, as the time from the first occurrence of response (CR or mCR or PR) to disease progression or death, whichever occurs first.
Progression Free Survival (PFS), for MDS | Up to approximately 3 years
  Progression Free Survival (PFS) defined as the time from the date of the first dose of any study drug to PD or death from any cause.
OS, for MDS | Up to approximately 3 years
  OS, defined as the time from the date of the first dose of any study drug to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (29):
- United States (9):
  - University of Alabama at Birmingham - Main /ID# 227071, Birmingham, Alabama
  - Norton Cancer Institute - St Matthews /ID# 228378, Louisville, Kentucky
  - Massachusetts General Hospital /ID# 227273, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 231083, Boston, Massachusetts
  - University of Michigan /ID# 227030, Ann Arbor, Michigan
  - University of Pennsylvania /ID# 227024, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Ctr /ID# 228048, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center at Texas Medical Center /ID# 227019, Houston, Texas
  - University of Virginia Health /ID# 227363, Charlottesville, Virginia
- Australia (2):
  - Liverpool Hospital /ID# 227723, Liverpool, New South Wales
  - Austin Health /ID# 227717, Heidelberg, Victoria
- Germany (4):
  - Marien Hospital Duesseldorf /ID# 227751, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 227750, Leipzig, Saxony
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 227749, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 227748, Hamburg
- Israel (4):
  - Hadassah Medical Center-Hebrew University /ID# 227275, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 227389, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 227387, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 227738, Petah Tikva
- Italy (3):
  - Istituto Clinico Humanitas /ID# 226948, Rozzano, Milano
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 226950, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 226952, Milan
- Japan (4):
  - National Cancer Center Hospital East /ID# 232498, Kashiwa-shi, Chiba
  - University of Fukui Hospital /ID# 232466, Yoshida-gun, Fukui
  - Kyushu University Hospital /ID# 232564, Fukuoka, Fukuoka
  - Yamagata University Hospital /ID# 232451, Yamagata, Yamagata
- Spain (3):
  - Hospital Clinic de Barcelona /ID# 227772, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 227771, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 227770, Málaga

IPD SHARING:
Plan to Share IPD: No